CLINICAL TRIAL: NCT05168761
Title: Complications Associated With Partial Nephrectomy for Renal Cancer: PMSI French National Data
Brief Title: Complications Associated With Partial Nephrectomy for Renal Cancer
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, ESCHWEGE Pascal, Professor, Central Hospital, Nancy, France
Other Study IDs: 2040/1205
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Renal Cancer; Partial Nephrectomy
Keywords: nephron sparing; robot; PMSI; laparoscopy; open surgery; nephron sparing surgery
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- laparoscopic partial nephrectomy: The investigators included all hospitalisations for LPN using CCAM(Classification Commune des actes médicaux) code (JAFC005) after removing the 83 hospitals using RAPN in 2017. LPN complications were from hospitals using exclusively LPN.
  Interventions: Procedure: partial nephrectomy
- open partial nephrectomy: OPN has its own CCAM codes; they group laparotomy (JAFA019 / JAFA030) and lumbotomy (JAFA008 / JAFA024)
  Interventions: Procedure: partial nephrectomy
- robot assisted partial nephrectomy: At the time of this study, RAPN did not have a specific coding. The investigators had contacted the hospitals with Vinci robotic surgical procedures in 2013 and the investigators included here PN from hospitalisations from the 25 centres using exclusively RAPN for more than five years. Thus, in this study, RAPN was performed by experts in robotic surgery.
  Interventions: Procedure: partial nephrectomy

INTERVENTIONS:
Procedure: partial nephrectomy

SUMMARY:
This paper evaluates the initial complications and the complications two years postoperatively necessitating re-hospitalisation for three surgical procedures for renal tumour partial nephrectomy .

DETAILED DESCRIPTION:
This paper evaluates the initial complications and the complications two years postoperatively necessitating re-hospitalisation for three surgical procedures for renal tumour partial nephrectomy (open (OPN), standard laparoscopy (LPN) and robot assisted laparoscopy (RAPN)) in 2016-2017 in France (9119 initial hospitalisations included 4035 OPN, 1900 RAPN, 1709 LPN). The investigators have extracted for these all hospitalisations from the French national hospital data base (PMSI-MCO). The investigators concluded mini-invasive and robotic surgery had lower morbidity and a shorter initial hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* hospitalisations between the 1st January 2016 and the 31st December 2017 with one of the partial nephrectomy codes

Exclusion Criteria:

* partial nephrectomy for non-cancerous pathology
* no technical information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In total, there were 11,698 hospitalisations between the 1st January 2016 and the 31st December 2017 with one of the PN codes from the Classification Commune des Actes Médicaux (CCAM) (Annex 1). The investigators used a supplementary filter for the diagnosis of renal cancer, C64, from the International Classification of Diseases 10th edition (ICD-10). The Department of Medical Informatics, Nancy CHRU controlled coding discrepancies, leaving 9119 hospitalisations for study
Sampling Method: Non-Probability Sample
Enrollment: 7664 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
post operative complication | 2 years
  Complications were documented for the initial hospitalisation and any subsequent re-hospitalisation

SECONDARY OUTCOMES:
length of initial hospitalisation | 2 years
  length of initial hospitalisation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungberg B, Albiges L, Abu-Ghanem Y, Bensalah K, Dabestani S, Fernandez-Pello S, Giles RH, Hofmann F, Hora M, Kuczyk MA, Kuusk T, Lam TB, Marconi L, Merseburger AS, Powles T, Staehler M, Tahbaz R, Volpe A, Bex A. European Association of Urology Guidelines on Renal Cell Carcinoma: The 2019 Update. Eur Urol. 2019 May;75(5):799-810. doi: 10.1016/j.eururo.2019.02.011. Epub 2019 Feb 23. PMID 30803729
- [Background] Hanzly M, Frederick A, Creighton T, Atwood K, Mehedint D, Kauffman EC, Kim HL, Schwaab T. Learning curves for robot-assisted and laparoscopic partial nephrectomy. J Endourol. 2015 Mar;29(3):297-303. doi: 10.1089/end.2014.0303. Epub 2014 Oct 21. PMID 25111313
- [Background] Gill IS, Kavoussi LR, Lane BR, Blute ML, Babineau D, Colombo JR Jr, Frank I, Permpongkosol S, Weight CJ, Kaouk JH, Kattan MW, Novick AC. Comparison of 1,800 laparoscopic and open partial nephrectomies for single renal tumors. J Urol. 2007 Jul;178(1):41-6. doi: 10.1016/j.juro.2007.03.038. Epub 2007 May 11. PMID 17574056
- [Background] Masson-Lecomte A, Bensalah K, Seringe E, Vaessen C, de la Taille A, Doumerc N, Rischmann P, Bruyere F, Soustelle L, Droupy S, Roupret M. A prospective comparison of surgical and pathological outcomes obtained after robot-assisted or pure laparoscopic partial nephrectomy in moderate to complex renal tumours: results from a French multicentre collaborative study. BJU Int. 2013 Feb;111(2):256-63. doi: 10.1111/j.1464-410X.2012.11528.x. Epub 2012 Dec 20. PMID 23279002
- [Background] Bravi CA, Larcher A, Capitanio U, Mari A, Antonelli A, Artibani W, Barale M, Bertini R, Bove P, Brunocilla E, Da Pozzo L, Di Maida F, Fiori C, Gontero P, Li Marzi V, Longo N, Mirone V, Montanari E, Porpiglia F, Schiavina R, Schips L, Simeone C, Siracusano S, Terrone C, Trombetta C, Volpe A, Montorsi F, Ficarra V, Carini M, Minervini A. Perioperative Outcomes of Open, Laparoscopic, and Robotic Partial Nephrectomy: A Prospective Multicenter Observational Study (The RECORd 2 Project). Eur Urol Focus. 2021 Mar;7(2):390-396. doi: 10.1016/j.euf.2019.10.013. Epub 2019 Nov 12. PMID 31727523
- [Background] Haute Autorité de Santé HAS. Évaluation de la néphrectomie totale ou partielle assistée par robot.; 2019. https://www.has-sante.fr/jcms/p_3103989/fr/evaluation-de-la-nephrectomie-totale-ou-partielle-assistee-par-robot
- [Background] Andersen MH, Mathisen L, Oyen O, Edwin B, Digernes R, Kvarstein G, Tonnessen TI, Wahl AK, Hanestad BR, Fosse E. Postoperative pain and convalescence in living kidney donors-laparoscopic versus open donor nephrectomy: a randomized study. Am J Transplant. 2006 Jun;6(6):1438-43. doi: 10.1111/j.1600-6143.2006.01301.x. PMID 16686768
- [Background] Camp C, O'Hara J, Hughes D, Adshead J. Short-term Outcomes and Costs Following Partial Nephrectomy in England: A Population-based Study. Eur Urol Focus. 2018 Jul;4(4):579-585. doi: 10.1016/j.euf.2017.03.010. Epub 2017 Apr 8. PMID 28753878
- [Background] Jain S, Nyirenda T, Yates J, Munver R. Incidence of renal artery pseudoaneurysm following open and minimally invasive partial nephrectomy: a systematic review and comparative analysis. J Urol. 2013 May;189(5):1643-8. doi: 10.1016/j.juro.2012.11.170. Epub 2012 Dec 3. PMID 23219544
- [Background] Peyronnet B, Seisen T, Oger E, Vaessen C, Grassano Y, Benoit T, Carrouget J, Pradere B, Khene Z, Giwerc A, Mathieu R, Beauval JB, Nouhaud FX, Bigot P, Doumerc N, Bernhard JC, Mejean A, Patard JJ, Shariat S, Roupret M, Bensalah K; French Comittee of Urologic Oncology (CCAFU). Comparison of 1800 Robotic and Open Partial Nephrectomies for Renal Tumors. Ann Surg Oncol. 2016 Dec;23(13):4277-4283. doi: 10.1245/s10434-016-5411-0. Epub 2016 Jul 13. PMID 27411552
- [Background] Zargar H, Khalifeh A, Autorino R, Akca O, Brandao LF, Laydner H, Krishnan J, Samarasekera D, Haber GP, Stein RJ, Kaouk JH. Urine leak in minimally invasive partial nephrectomy: analysis of risk factors and role of intraoperative ureteral catheterization. Int Braz J Urol. 2014 Nov-Dec;40(6):763-71. doi: 10.1590/S1677-5538.IBJU.2014.06.07. PMID 25615258
- [Background] Schmid M, Chiang HA, Sood A, Campbell L, Chun FK, Dalela D, Okwara J, Sammon JD, Kibel AS, Menon M, Fisch M, Trinh QD. Causes of hospital readmissions after urologic cancer surgery. Urol Oncol. 2016 May;34(5):236.e1-11. doi: 10.1016/j.urolonc.2015.11.019. Epub 2015 Dec 23. PMID 26712365
- [Background] Achit H, Guillemin F, Karam G, Ladriere M, Baumann C, Frimat L, Hosseini K, Hubert J. Cost-effectiveness of four living-donor nephrectomy techniques from a hospital perspective. Nephrol Dial Transplant. 2020 Nov 1;35(11):2004-2012. doi: 10.1093/ndt/gfz143. PMID 31377771
- [Background] Ficarra V, Novara G, Secco S, Macchi V, Porzionato A, De Caro R, Artibani W. Preoperative aspects and dimensions used for an anatomical (PADUA) classification of renal tumours in patients who are candidates for nephron-sparing surgery. Eur Urol. 2009 Nov;56(5):786-93. doi: 10.1016/j.eururo.2009.07.040. Epub 2009 Aug 4. PMID 19665284
- [Background] Patel HD, Mullins JK, Pierorazio PM, Jayram G, Cohen JE, Matlaga BR, Allaf ME. Trends in renal surgery: robotic technology is associated with increased use of partial nephrectomy. J Urol. 2013 Apr;189(4):1229-35. doi: 10.1016/j.juro.2012.10.024. Epub 2012 Oct 17. PMID 23085300
- [Background] Tikkinen KAO, Craigie S, Agarwal A, Violette PD, Novara G, Cartwright R, Naspro R, Siemieniuk RAC, Ali B, Eryuzlu L, Geraci J, Winkup J, Yoo D, Gould MK, Sandset PM, Guyatt GH. Procedure-specific Risks of Thrombosis and Bleeding in Urological Cancer Surgery: Systematic Review and Meta-analysis. Eur Urol. 2018 Feb;73(2):242-251. doi: 10.1016/j.eururo.2017.03.008. Epub 2017 Mar 23. PMID 28342641
- [Background] Georgescu I, Hartmann FG. Sources of financial pressure and up coding behavior in French public hospitals. Health Policy. 2013 May;110(2-3):156-63. doi: 10.1016/j.healthpol.2013.02.003. Epub 2013 Mar 9. PMID 23477807